CLINICAL TRIAL: NCT00004208
Title: Antithymocyte Globulin (ATG) and Cyclosporine (CSA) to Treat Patients With Myelodysplastic Syndrome (MDS). A Randomized Trial Comparing ATG + CSA With Best Supportive Care
Brief Title: Antithymocyte Globulin and Cyclosporine in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 33/99; SWS-SAKK-33/99 (Other: SAKK)
Record Dates: First submitted 2000-01-21; First posted 2003-01-27 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: ATG + CSA (Active Comparator): Treatment consists of 15 mg/kg ATG (Mérieux; horse antithymocyte globulin; i.e. 1.5 vial/10 kg of body weight/day) given over 8-12 hours for 5 consecutive days.
  Cyclosporine A (CSA) will be administered orally in a dose of 2.5 mg/kg bid starting day 1 and continued through day 180.
  Interventions: Drug: ATG + CSA
- Arm B: Supportive care (Other): Patients randomized to this arm will be treated as outpatients.
  Interventions: Behavioral: Supportive care

INTERVENTIONS:
Drug: ATG + CSA — Mérieux; horse antithymocyte globulin (ATG) + Cyclosporine A (CSA)
  Arms: Arm A: ATG + CSA
Behavioral: Supportive care — Patients randomized to this arm will be treated as outpatients.
  Arms: Arm B: Supportive care

SUMMARY:
The main objective of this trial is to evaluate the efficacy and toxicity of intensive immuno-suppression with ATG + CSA versus best supportive care in patients with transfusion dependent low and intermediate risk myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
This trial will answer the question whether immuno-suppression improves hematopoesis and reduces transfusion requirements analogous to patients with aplastic anemia as the short-term outcome, and whether immuno-suppression accelerates leukemic transformation and influences survival as the long-term outcome.

Primary endpoint: best response (CR + PR) rate at month 6

ELIGIBILITY:
Hypoplastic MDS, or MDS subtype RA, RAS or RAEB with ≤ 10% blasts, or RAEB with 10-20% blasts and the patient refusing or not eligible for the MDS high risk protocol (EORTC 06961)

* Transfusion dependence < 24 months or neutrophils < 0.5 × 109/l.
* ECOG/SAKK performance status ≤ 2
* Age > 18 years
* No active uncontrolled infection
* No prior chemotherapy or radiotherapy
* No history of heart failure, clinically relevant cardiac arrhythmia or other hemato-oncological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2000-08; Primary Completion 2006-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Best response rate (CR + PR) | 6 months

SECONDARY OUTCOMES:
Response rate at month 3, time to response, quality and duration of response, and proportions of relapse/progression in responders | 2 and 5 years after first response
Overall survival | 2 and 5 years
Leukemia-free survival | 2 and 5 years
Transformation-free survival | 2 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jakob R. Passweg, MS, Study Chair — Kantonsspital Basel
Locations (1):
- Universitaetsspital-Basel, Basel, Switzerland

REFERENCES:
- [Result] Passweg JR, Giagounidis AA, Simcock M, Aul C, Dobbelstein C, Stadler M, Ossenkoppele G, Hofmann WK, Schilling K, Tichelli A, Ganser A. Immunosuppressive therapy for patients with myelodysplastic syndrome: a prospective randomized multicenter phase III trial comparing antithymocyte globulin plus cyclosporine with best supportive care--SAKK 33/99. J Clin Oncol. 2011 Jan 20;29(3):303-9. doi: 10.1200/JCO.2010.31.2686. Epub 2010 Dec 13. PMID 21149672
- [Result] Passweg JR, Giagounidis A, Simcock M, et al.: Immunosuppression for patients with low and intermediate risk myelodysplastic syndrome: a prospective randomized multicenter trial comparing antithymocyte globulin + cyclosporine with best supportive care: SAKK 33/99. [Abstract] Blood 110 (11): A-1461, 2007.